CLINICAL TRIAL: NCT03565081
Title: Effects of Progressive Elastic Band Resistance Training on Body Composition and Motor Performance in Adults With Prader-Willi Syndrome: a Pilot Study
Brief Title: Effects of Progressive Elastic Band Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-XD33-100
Record Dates: First submitted 2018-05-28; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-05

CONDITIONS: Prader-Willi Syndrome; Resistance Training
Keywords: Prader-Willi Syndrome; Resistance Training; Body Composition
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PWS elastic band training group (Experimental): Genetically confirmed diagnosis of PWS participants were recruited. The PWS participants needed to have sufficient command of the Mandarin language to understand the study information and motivated to conduct the training program.
  Interventions: Device: PWS elastic band training group

INTERVENTIONS:
Device: PWS elastic band training group — PWS participants received 9 sets exercises for the major muscle groups, over 24 weeks, three times a week, for a total of 72 sessions.

SUMMARY:
Abnormal body composition with increased body fat mass and decreased lean body mass has been found in adults with Prader-Willi syndrome (PWS), contributing to reduced physical capacity and impairment. The aim of this study was to investigate whether progressive elastic band resistance training can improve physical motor performance and regional body composition in adults with PWS.

DETAILED DESCRIPTION:
Six participants were enrolled in this pilot study. Following 24 weeks of progressive elastic band resistance exercise training, significant reduction was observed in their body weight, BMI, and regional extremities fat mass and percentage. Regarding the functional performances, there were also significant improvements in their hand grip strength, 3 meter timed up and go, 30 seconds sit to stand, and 2-min step up tests, as early as the 8th week of training. Balance function achieved significant improvements after 16 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* PWS individuals who can cooperate with motor performances

Exclusion Criteria:

* arthritis, fracture, or severe musculoskeletal deformities that would interfere with exercise training or motor performance
* severe cognitive impairment or parents who cannot read nor write.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in the handgrip strength functional physical assessment | Changes from Baseline functional motor performance tests at 8 weeks, 16 weeks and 24 weeks
  hand grip strength (pounds),
Changes in the 30 second chair stand functional physical assessment | Changes from Baseline functional motor performance tests at 8 weeks, 16 weeks and 24 weeks
  30-second chair stand test (times)
Changes in the timed up and go functional physical assessment | Changes from Baseline functional motor performance tests at 8 weeks, 16 weeks and 24 weeks
  timed up-and-go test (seconds)
Changes in the two minute step up functional physical assessment | Changes from Baseline functional motor performance tests at 8 weeks, 16 weeks and 24 weeks
  2 minute step up test (times)
Changes in the balance functional physical assessment | Changes from Baseline functional motor performance tests at 8 weeks, 16 weeks and 24 weeks
  Berg Balance Scale (0-56 points; 0-20= high fall risk; 21-40= medium fall risk; 41-56= low fall risk)
Change in the BMI body composition | Change from Baseline body composition components at 6 months
  Body weight (km) and height (m) will be combined to report as BMI (kg/m2)
Change in the percentage of body fat of body composition | Change from Baseline body composition components at 6 months
  Regional percentage body fat (%)
Change in the body fat mass of body composition | Change from Baseline body composition components at 6 months
  Fat mass (kg)
Change in the lean body mass of body composition | Change from Baseline body composition components at 6 months
  Lean body mass (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Valeria JY Chiu, MD, Principal Investigator — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Foundation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schlumpf M, Eiholzer U, Gygax M, Schmid S, van der Sluis I, l'Allemand D. A daily comprehensive muscle training programme increases lean mass and spontaneous activity in children with Prader-Willi syndrome after 6 months. J Pediatr Endocrinol Metab. 2006 Jan;19(1):65-74. doi: 10.1515/jpem.2006.19.1.65. PMID 16509530
- [Result] Eiholzer U, Nordmann Y, l'Allemand D, Schlumpf M, Schmid S, Kromeyer-Hauschild K. Improving body composition and physical activity in Prader-Willi Syndrome. J Pediatr. 2003 Jan;142(1):73-8. doi: 10.1067/mpd.2003.mpd0334. PMID 12520259